CLINICAL TRIAL: NCT03586336
Title: Remote Dielectric Sensing Technology Guided Diuresis in Hospitalized Patients With Acute Decompensated Heart Failure
Brief Title: Remote Dielectric Sensing (ReDS) Assisted Diuresis in Acute Decompensated Heart Failure
Acronym: RADAR-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Sensible Medical Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RADAR-HF
Record Dates: First submitted 2018-06-13; First posted 2018-07-13 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; With Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ReDS-Guided (Experimental): Patients in the intervention arm will undergo daily measurements of lung fluid content at the bedside with the ReDS vest. The values will be shared with the treating clinicians, who can use the measurements in addition to other standard data to guide diuresis. Patients should be discharged only once their lung fluid content falls within the normal range of 20-35%.
  Interventions: Device: ReDS-Guided
- Control (Sham Comparator): Patients in the control arm will also undergo daily measurements of lung fluid content at the beside with the ReDS vest. However, the values will not be shared with the treating clinicians, who will direct management based on standard clinical tools
  Interventions: Device: Usual Care

INTERVENTIONS:
Device: ReDS-Guided — ReDS measurements will be shared with the treating clinicians who can use the information to guide diuresis and determine the appropriate timing of discharge
  Arms: ReDS-Guided
Device: Usual Care — ReDS measurements will not be shared with the treating clinicians, who will guide diuresis using standard clinical criteria
  Arms: Control

SUMMARY:
This study evaluates the use of a wearable vest capable of non-invasively measuring lung fluid content in hospitalized patients with heart failure

DETAILED DESCRIPTION:
Inpatient management of acute decompensated heart failure centers around the efficient relief of congestion with IV diuretics and vasoactive agents. For the majority of patients, non-invasive, clinical bedside tools such as jugular venous pressure, pulmonary auscultation and daily weights are used to estimate cardiac filling pressures and guide diuresis. However, these methods are subject to significant inter-observer variability and can be unreliable for various reasons. Furthermore, recent studies have shown that overt signs of clinical congestion correlate poorly with hemodynamic congestion assessed by invasive means. Remote Dielectric Sensing is a novel technology that enables the non-invasive assessment of lung fluid content using a wearable vest. ReDS measurements have been shown to correlate with fluid status in hospitalized HF patients and have been used to remotely monitor ambulatory HF patients for signs of pre-clinical hemodynamic congestion. In this prospective, randomized study, we will assess the utility of ReDS guided diuresis in hospitalized patients with acute decompensated heart failure. All patients will receive daily ReDS measurements, but only treating physicians in the intervention group will be able to use these values to guide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for acute decompensated heart failure requiring treatment with intravenous diuretics and/or IV vasoactive drugs
* Patient has signed informed consent and has authorized use and disclosed health information
* Patient is at least 18 years of age
* Patient physically suitable for ReDS measurement
* GFR>25
* Initial ReDS Measurement >35%

Exclusion Criteria:

* Patient characteristics excluded from approved use of ReDS system: height less than 155cm or greater than 190cm, BMI <22 or >39, chest circumference <80cm or >115cm , or flail chest
* Evidence of focal lung lesions on history, physical exam or chest x-ray, including history of pulmonary embolism, active pneumonia, or known lung nodule
* Chronic renal failure (GFR<25)
* Prior cardiac surgery within 2 months of index admission
* Patient has a ventricular assist device or has had a cardiac transplantation
* Patients in cardiogenic shock at admission requiring inotropic support
* Congenital heart malformations or intra-thoracic mass that would affect right-lung anatomy (e.g dextrocardia, lung carcinoma, or pacemaker box in the right chest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Net Fluid Balance during hospitalization | During hospitalization, approximately 7 days
  Cumulative net fluid balance assessed by In's and Out's recorded in the Electronic Medical Record (EMR) during hospitalization

SECONDARY OUTCOMES:
Change in GFR from admission to discharge | During hospitalization, approximately 7 days
  Net change in GFR (calculated using the Chronic Kidney Disease Epidemiology 2009 equation) from admission to discharge
Length of Stay in hospital | During hospitalization, approximately 7 days
  Duration of hospitalization
Major adverse cardiac events at 30 days | 30 Days after discharge
  The combined rate of cardiovascular mortality or heart failure readmission at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Liviu Klein, MD, MS, Principal Investigator — Director, Mechanical Circulatory Support and Heart Failure Device Program
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gheorghiade M, Pang PS. Acute heart failure syndromes. J Am Coll Cardiol. 2009 Feb 17;53(7):557-573. doi: 10.1016/j.jacc.2008.10.041. PMID 19215829
- [Background] Amir O, Ben-Gal T, Weinstein JM, Schliamser J, Burkhoff D, Abbo A, Abraham WT. Evaluation of remote dielectric sensing (ReDS) technology-guided therapy for decreasing heart failure re-hospitalizations. Int J Cardiol. 2017 Aug 1;240:279-284. doi: 10.1016/j.ijcard.2017.02.120. Epub 2017 Mar 3. PMID 28341372
- [Background] Amir O, Rappaport D, Zafrir B, Abraham WT. A novel approach to monitoring pulmonary congestion in heart failure: initial animal and clinical experiences using remote dielectric sensing technology. Congest Heart Fail. 2013 May-Jun;19(3):149-55. doi: 10.1111/chf.12021. Epub 2013 Jan 25. PMID 23350643